CLINICAL TRIAL: NCT01336114
Title: A New 3D Geometrical Modelisation of Adolescent Idiopathic Scoliosis and Conception of a Personal Brace
Acronym: MODEL MAKER
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-A01263-36; LOC/10-14
Record Dates: First submitted 2011-04-06; First posted 2011-04-15 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Adolescent idiopathic scoliosis (AIS) involves complex tridimensional deformities of the spine. In case of progressive curve deformity, the use of spinal bracing remains the standard non operative treatment of moderate AIS. Most of the time, the different types of braces don't take into account the individual biomechanical properties of each patient's spine. Actually, it is essential to better understand the effect of the loads applied on the trunk and on the spine, and a 3D geometrical modelisation of these components is essential. Many studies have been publishing concerning the use of radiographs for the geometrical reconstruction of the spine, and more recently the EOS system. But even then, it is still necessary to obtain an important number of geometrical data and discretisation is still a long procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* Pre menarchial for the girls
* Risser 0 et Risser 3 on X rays. Radiologic classification of spine maturity (ossification of the iliac crests). Five stages.
* Cobb angle ≥25° and < 40°
* Information to the parents and child, and signed approval

Exclusion Criteria:

* No idiopathic scoliosis
* Previous brace treatment
* Immediate indication for surgery
* Previous thoracic surgery

Ages: 12 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with idiopathic scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-07

PRIMARY OUTCOMES:
Photographs of the back and spine radiographs for making a corset | 3 years
  The torso shape reconstruction is realized thanks to the system Model Maker(Proteor®) on adolescent idiopathic patients. Model Maker allows to reconstruct the external shape of the human body from about 20 images steaming from a standard digital camera.The spine reconstruction is has for her obtained by means of a software interface, from tow standard clinical X-rays in the digital format (frontal and sagittal) and images were used by Model Maker for the external shape reconstruction.

SECONDARY OUTCOMES:
Recording of pressure from the brace | 3 years
  The recording of pressure from the brace is done through a web of pressure positioned in the brace. It is a structure "teck scan (Expert-Seat, Ergoresearch Inc)" containing polymeric pressure sensors. The pressure exerted by the brace on the trunk is registered in different positions (standing, lying).

CONTACTS AND LOCATIONS:
Overall Officials: philippe violas, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France